CLINICAL TRIAL: NCT05413876
Title: Fabry Exercise Intolerance Study (FEISTY)
Brief Title: Fabry Exercise Intolerance Study
Acronym: FEISTY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Dr. Mirjam Langeveld, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL73534.018.21
Record Dates: First submitted 2022-05-17; First posted 2022-06-10 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Fabry Disease; Fabry Disease, Cardiac Variant
MeSH Terms: conditions — Fabry Disease; Fabry Disease, Cardiac Variant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Men with classical Fabry disease
  Interventions: Other: Intermittent cardiopulmonary exercise test; Other: Incremental cardiopulmonary exercise test
- Women with classical Fabry disease
  Interventions: Other: Intermittent cardiopulmonary exercise test; Other: Incremental cardiopulmonary exercise test
- Men with non-classical Fabry disease
  Interventions: Other: Intermittent cardiopulmonary exercise test; Other: Incremental cardiopulmonary exercise test
- Healthy controls: Age-, Sex-, BMI-matched controls
  Interventions: Other: Intermittent cardiopulmonary exercise test; Other: Incremental cardiopulmonary exercise test

INTERVENTIONS:
Other: Intermittent cardiopulmonary exercise test — Exercise test with step-change from rest to a relatively low constant workload.
Other: Incremental cardiopulmonary exercise test — Exercise test with incremental workload until maximal workload.

SUMMARY:
Patients and healthy controls will undergo cardiopulmonary exercises and testing of the muscles strength to gain additional understanding of exercise intolerance as Fabry disease (FD) manifestation. An additional needle muscle biopsy may be performed. Tissue analysis from this biopsy will include evaluation of the lipidomics profile and mitochondrial function. Results of the tests and any potential exercise intolerance will be compared against healthy, age-, sex- and BMI-matched volunteers. The hypothesis is that patients with FD will have reduced exercise capacity due to changes in skeletal and cardiac muscle energy metabolism.

DETAILED DESCRIPTION:
Background: Fabry disease (FD) is an inherited, highly variable and slowly progressive X linked disorder, which predominantly affects vascular endothelium, the heart, kidneys and the brain. Exercise intolerance is a complaint expressed by the majority of patients, at all stages of the disease. The exact cause, extent and development over time of exercise intolerance in FD in insufficiently understood. This limits preventive measures and adequate treatment.

Hypothesis: 1) The development of energy metabolism in skeletal and cardiac muscle in FD is disturbed early on in disease development and this progresses as the disease worsens, resulting in reduced exercise capacity. 2) Intermittent CPX is an objective and sensitive tool to grade the level of exercise tolerance in FD patients and yields specific outcome parameters that can be used in future intervention studies.

Primary objectives: 1) To study the presence and extent of exercise intolerance in male, female FD patients with classical FD and men with non-classical FD, in different stages of the disease. 2) To determine the aetiology of exercise intolerance in FD. Secondary objectives: 1) To determine whether the exercise test protocol used in this study can be used as a clinical outcome measure in future intervention studies. 2) To investigate difference in the time-relation between V'O2 and circulatory, ventilatory and metabolic variables during intermittent exercise between FD patients groups (potentially providing an indication of the source of possibly slowed V'O2 kinetics).

Methods: This study will consist of two screening visits, one testing procedure visit, and an optional second visit for all subjects enrolled in the study. During the first testing visit two cardiopulmonary exercise (CPX) test will be performed. During the CPX tests gas exchange, ventilation, blood pressure and cardiac output will be measured and exhaustion level monitored. Before and after the tests a blood sample will be taken. The upper leg muscle strength and the leg muscle size will be assessed. In order to detect alterations in skeletal muscle energy metabolism, a needle biopsy of the upper leg muscle will be taken during the second optional study visit. In the biopsy specimen, lipidomics profile, electronic microscopic characteristics of muscle tissue and mitochondrial function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* FD patients: Men and women with a definite known diagnosis of FD.
* Healthy controls: Healthy control subjects (men and women) with an age of 18 years of older.

Exclusion Criteria:

FD patients:

* Pregnancy
* Recent acute myocardial infarct (<6 months)
* Uncontrolled arrhythmia/severe conduction disorder (atrial fibrillation or second/third-degree AV block) causing hemodynamic compromise
* Implantable pacemaker or other cardiac device with complete ventricular pacing
* Uncontrolled heart failure with hemodynamic compromise
* Uncontrolled hypertension (Systolic Blood Pressure >150 mmHg and Diastolic Blood Pressure >100 mmHg on repeated measurements)
* Active infection, anaemia, severe renal dysfunction (estimated Glomerular filtration rate <30 ml/min/1,73m2) likely to significantly impact on exercise performance
* In some cases: use of anticoagulants or anti platelet therapy (see study procedure)

Healthy controls:

* All abovementioned exclusion criteria for FD patients
* History of smoking
* History of active drug use which can affect exercise intolerance
* History of asthma, chronic obstructive pulmonary disease, heart failure, heart surgery, heart rhythm disorders or congenital heart diseases
* Use of chronic medication likely to affect exercise tolerance
* Chronic illness (including orthopaedic, endocrinological, haematological, malignant, gastrointestinal, neurological, muscle or inflammatory disorders) likely to significantly impact on exercise performance
* >6 alcohol units per day or >14 alcohol units per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population of FD patients, either with a classical or a non-classical phenotype.
  Population of healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2024-01-02 (Estimated); Study Completion 2024-01-02 (Estimated)

PRIMARY OUTCOMES:
Differences in V'O2 max kinetics (ml/kg/min) | At rest (baseline) and after maximum CPX test (30 min)
Tiffeneau-index (FEV1/IVC ratio) | At rest (baseline)
  Pulmonary involvement
Anaerobic threshold (ml/kg/min) | During maximum exercise (max 30 min).
  Pulmonary involvement/Cardiac dysfunction/Skeletal muscle alterations
Ventilation reserve (L) | During maximum exercise (max 30 min).
  Pulmonary involvement/Skeletal muscle alterations
CO2 ventilation equivalent (L/L) | During maximum exercise (max 30 min).
  Pulmonary involvement/Cardiac dysfunction
O2 saturation (%) | During maximum exercise (max 30 min).
  Pulmonary involvement/Cardiac dysfunction
Cardiac Output (L/min) | During maximum exercise (max 30 min).
  Cardiac dysfunction
Heart rate reserve (per minute) | During maximum exercise (max 30 min).
  Cardiac dysfunction:
Muscle size on echography (cm) | Baseline
  Skeletal muscle alterations
Muscle strength via resistance test (kg) | Biopsy at baseline
  Skeletal muscle alterations
Lipidomics profile of muscle tissue | Biopsy at baseline
  Skeletal muscle alterations
Electronic microscopic characteristics of muscle tissue | Biopsy at baseline
  Skeletal muscle alterations
Mitochondrial function of muscle tissue | Biopsy at baseline
  Skeletal muscle alterations

SECONDARY OUTCOMES:
Correlation between V'O2 kinetics during intermittent exercise and V'O2 max on the incremental maximum CPX (Pearson correlation coefficient). | Day 1
Correlation between V'O2 kinetics during intermittent exercise and activity score on the SQUASH Questionnaire (Pearson correlation coefficient). | Day 1
Correlation between V'O2 kinetics during intermittent exercise and functional and morphological cardiac parameters on cardiac imaging (Magnetic resonance or echocardiography) (Pearson correlation coefficient). | Day 1

OTHER OUTCOMES:
Body height (cm) | Baseline
Body weight (kg) | Baseline
NT-proBNP (ng/L) | Baseline
Troponin (μg/L) | Baseline
Lactate (mmol/L) | Baseline and after maximum exercise
Haemoglobin (mmol/L) | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands